CLINICAL TRIAL: NCT00805805
Title: Phase III Trial of Tetrathiomolybdate (TM) in Primary Biliary Cirrhosis
Brief Title: Study Comparing Tetrathiomolybdate vs Standard Treatment in Primary Biliary Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: George Brewer (Other)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, George Brewer, Professor, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBC
Record Dates: First submitted 2008-12-08; First posted 2008-12-10 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Primary Biliary Cirrhosis
Keywords: Copper; ceruloplasmin; tetrathiomolybdate
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — tetrathiomolybdate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Tetrathiomolybdate with ursodiol
  Interventions: Drug: Tetrathiomolybdate
- 2 (Placebo Comparator): Placebo with ursodiol
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tetrathiomolybdate — 120 mg/day, divided as 20 mg three times/day with meals and 60 mg away from food at bedtime, for one week to test gastric tolerance. Increased to 180 mg/day, divided as 40 mg three times/day with meals and 60 mg away from food at bedtime. Serum ceruloplasmin levels measured weekly will be used as a surrogate measure of copper status, with a target of 10-15 mg/dl (normal 20-40). When target Cp levels are reached, usually in 4-8 weeks, a maintenance dose of usually 40-80 mg of TM/day, divided half with a major meal, and half away from food at bedtime will be established (vary from 10 mg to 120 mg/day).
  Arms: 1
Other: Placebo — Arm 2 will basically mirror Arm 1 with the patients receiving 120 mg/day, divided as 20 mg three times/day with meals and 60 mg away from food at bedtime the first week. Increased to 180 mg/day, divided as 40 mg three times/day with meals and 60 mg away from food at bedtime. With the dosage being reduced at about the same frequency as the patients receiving TM
  Arms: 2

SUMMARY:
The University of Michigan is conducting a study investigating a potential new treatment aimed at slowing/halting progression of primary biliary cirrhosis. This will be a 2 arm double blind study in which half of the patients will be randomly selected to receive a placebo (capsule with no active ingredient) and half will receive the new treatment drug, tetrathiomolybdate. Neither the patient nor the treating physician will know which arm the patient is in. The length of the study for each patient is 24 months of drug therapy. Lab draws will be necessary weekly for the first 6 weeks of the study, followed by every other week for 3 weeks, and then monthly for the remainder of the 2 year period. In addition, intermittent history and physicals and urine samples will also be necessary. There is no cost to you for any experimental treatment. All patients in both arms will continue on ursodiol and receive standard of care treatment

ELIGIBILITY:
Inclusion Criteria:

* Generally medically healthy
* Age 18 and older
* Documented primary biliary cirrhosis
* Alkaline phosphatase > 137

Exclusion Criteria:

* Severe liver decompensation
* Requirement for renal dialysis
* Pregnancy or nursing
* Meld score > 15 (13-15 will require a physician's clinical judgment)
* Uncontrolled congestive heart failure
* Severe diabetic neuropathy
* Severe pulmonary disease
* Advanced cancer
* Requirement for steroid therapy
* Uncontrolled ascites, variceal hemorrhage or spontaneous bacterial peritonitis
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Improvement in drug treated group vs placebo group in two liver function tests and one serum cytokine measurement | 2 years

SECONDARY OUTCOMES:
Improvement in drug treated group vs placebo group in serum CRP or interleukin-1-beta-levels | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States